CLINICAL TRIAL: NCT04034602
Title: Immediate Effect of Plantar Vibration on Fall Risk and Postural Stability in Stroke Patients
Brief Title: Immediate Effect of Plantar Vibration on Fall Risk and Postural Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Birol Önal, research assistant, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: vibrationimmediateeffect
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Stroke Patients
Keywords: stroke vibration fall risk postural stability; immediate effect; fall risk; postural stability

STUDY DESIGN:
Intervention Model Description: 30 stroke patients will be included in this study. The patients who meet the inclusion criteria will be divided randomly into 2 groups as vibration (n=15) and placebo (n=15).The vibration group, one session in supine position will be applied to both sides of the soles of the feet under the soles of the feet for 5 minutes with a 15-100 Hz frequency CE certified vibration device. In the placebo group, both sides will be held in the supine position under the soles of the foot for 5 minutes each so that the device is in contact with the foot without vibration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vibration group (Experimental): plantar vibration group is supine position, plantar vibration will be applied to both foot of each patient with a vibration device with a frequency of 15-100 Hz over 5 minutes.
  Interventions: Other: vibration group
- placebo group (Active Comparator): the placebo group, both sides will be held in the supine position under the soles of the foot for 5 minutes each so that the device is in contact with the foot without vibration.
  Interventions: Other: placebo group

INTERVENTIONS:
Other: vibration group — plantar vibration group is supine position, plantar vibration will be applied to both foot of each patient with a vibration device with a frequency of 15-100 Hz over 5 minutes.
  Arms: vibration group
Other: placebo group — the placebo group, both sides will be held in the supine position under the soles of the foot for 5 minutes each so that the device is in contact with the foot without vibration.
  Arms: placebo group

SUMMARY:
The aim of this study; To determine the immediate effect on fall risk and postural stability of vibration applied to the plantar region in stroke patients.

DETAILED DESCRIPTION:
Kırıkkale University Faculty of Medicine Physical Therapy will be hospitalized in the USA clinic and volunteers will be involved in stroke rehabilitation. The patients who meet the inclusion criteria and who are excluded from the exclusion criteria will be randomized according to the order of arrival and will be divided into two groups as the vibration group and the placebo group.Patients will be taken to the placebo and vibration group respectively in order of arrival. If the next patient falls outside the inclusion criteria of the study, randomization will be applied to the next patient. The vibration group, one session in supine position will be applied to both sides of the soles of the feet under the soles of the feet for 5 minutes with a 15-100 Hz frequency CE certified vibration device. In the placebo group, both sides will be held in the supine position under the soles of the foot for 5 minutes each so that the device is in contact with the foot without vibration.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive and non-communication problems
* Volunteer to join the work
* Those with less than 150 kilos
* Spasticity according to a Modified Scale Ashworth 2 and 3 patients treated with Botox
* Patients at least 8 weeks after stroke diagnosis

Exclusion Criteria:

* People who are not stable due to vital signs
* Open wounds under the soles of the feet
* Being spastic at the level that will block the base touch
* Pathological conditions affecting lower limb sense (diabetic peripheral neuropathy, post- fracture surgery)
* 20 seconds independent standing
* Mini Mental Test score below 24
* Multiple sclerosis, Parkinson's disease, etc.
* Those with vision problems
* Patients with thoracolumbar surgery
* Patients with spinal canal stenosis

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
biodex balance system fall risk test | 5 minutes
  Fall Risk Test is a test used to determine the risk of falling. The higher the score, the higher the risk of falling. The device compares the test results with normal age-related data to calculate the risk of falling, the platform was set to move from 12 to 8, with the platform moving. The test is carry out with 3 repetitions, each with a resting time of 10 seconds each, lasting 20 's each while the platform is static. On the support surface formed by placing the two legs in a comfortable position on the platform, it is requested to keep the black dot on the screen of the device in the middle of the visual on the screen for 20 seconds. The average of these 3 repetitions is automatically calculated by the device for the risk of falling.
biodex balance system postural stability test | 5 minutes
  The Postural Stability Test assessment the participant's ability to control the center of gravity. The extent to which the participant's position deviates from the center is measured and reports the mean deviation as the stability index. A low score indicates that the amount of deviation is small and postural stability is good. If the standard deviation is high, the participant's postural oscillation is also high when the test platform is in a static state, each is 20 seconds lasting, between 10 seconds rest period was done as 3 repetitions. On the support surface formed by placing the two legs in a comfortable position on the platform, it was requested to keep the black dot on the screen of the device in the middle of the visual on the screen for 20 seconds. For the Mediolateral Stability Index, Anterioposterior Stability Index and General Stability Index showing the postural stability, the mean of 3 replicates of this test was automatically calculated by the device.

CONTACTS AND LOCATIONS:
Overall Officials: Birol Önal, Principal Investigator — Kirikkale Univercity
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No